CLINICAL TRIAL: NCT05915117
Title: Randomized, Double-blind, Placebo-controlled Study of Efficacy Polyphenols of Pomegranate Fruit Peel Extract on Inflammatory Parameters and Oxidative Stress in Overweight and Obese Subjects With Metabolic Syndrome
Brief Title: Effects of Polyphenols of Pomegranate Fruit Peel Extract on Inflammation and Oxidative Stress in Metabolic Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Banja Luka (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PoPexMetSy
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-04

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic syndrome; Inflamation; Oxidative stress; Obesity; Polyphenols of Pomegranate Fruit Peel Extract
MeSH Terms: conditions — Metabolic Syndrome; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polyphenols of pomegranate fruit peel extract (PoPex) (Experimental): All subjects will treated only with PoPex in total daily dosis of 500 mg/orally over 8 weeks.
  Interventions: Dietary Supplement: Polyphenols of pomegranate fruit peel extract (PoPex)
- Placebo (Placebo Comparator): All subjects will treated only with PoPex placebo capsules/orally over 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Polyphenols of pomegranate fruit peel extract (PoPex) — PoPex in form of capsule will be orally administered in total daily dose of 500/mg in subjects with metabolic syndrome and obesity over 8 weeks.
  Other Names: Granat
  Arms: Polyphenols of pomegranate fruit peel extract (PoPex)
Drug: Placebo — Placebo in form of capsule will be orally administered in subjects with metabolic syndrome and obesity over 8 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effects of polyphenols of pomegranate fruit peel extract compared to placebo on oxidative stress and inflammation in overweight and obese subjects with metabolic syndrome.

DETAILED DESCRIPTION:
This is a Phase 3, randomized, double-blind, placebo-controlled evaluation of the efficacy of polyphenols of pomegranate fruit peel extract on oxidative stress and inflammation in overweight and obese subjects with metabolic syndrome.

Study site: a single study center (Primary Health Care Institution in Banja Luka, as recruiter center) as recruitment center including Center for Biomedical Research, Faculty of Medicine University of Banja Luka, as local laboratory and coordinator.

Sample size: 60 subjects, randomized in a 1:1 allocation ratio.

Primary objectives are to investigate an effect of polyphenols pomegranate fruit peel extract on: Anthropometric parameters such as body mass index, and arterial blood pressure, glycemia, lipoprotein profile, homeostatic model assessment for insulin resistance (HOMAIR), homocysteine, vitamin B complex: folic acid, vitamin B6, vitamin B9 and vitamin B12.

2. To investigate the effects polyphenols from pomegranate fruit peel extract has on impact on lipid peroxidation index, nitric oxide metabolites, hydrogen peroxide (H2O2), superoxide anion radical (O2-), and glutathione (GSH), catalase (CAT) and superoxide dismutase (SOD).

3. Proinflammatory markers interleukin-6 (IL-6), tumor necrosis factor-α (TNF-α), high sensitive CRP (hsCRP), leptin, resistin ,vaspin, chemerin, lipokalin-2 and katepsin .

4. Anti-infammatory markers IL-5, IL-10, IL-12 ,adiponectin and omentin.

Treatments arms:

Polyphenols of pomegranate fruit peel extract (PoPeEx) (500 mg/day) Placebo

Treatment duration :

8 weeks

Assessment - clinical and laboratory sampling:

Informed consent and Screening - 7 days prior to randomization

Study visits (V):

V1 - Randomization and Enrollment (Baseline) V2 - 4 weeks after Baseline V3 - 8 weeks after Baseline.

No interim analysis is planned. The analysis will be performed at the end of the study after data review and freezing of the database according to the intent to treat principle.

- Page 2 of 6 [DRAFT] -

ELIGIBILITY:
Inclusion Criteria:

Informed consent signed Adults of 20 to 60 years BMI ≥ 25.00 kg/m2

Met criteria for metabolic syndrome such as visceral obesity( for men ≥ 94 cm and ≥ 80 cm for women) and at least two risk factors:

1. TG ≥ 1,7 mmol/l, or present therapy for dyslipidemia
2. HDL <1,03 mmol/l men, <1,29 mmol/l women
3. Arterial blood pressure ≥130/85 mmHg
4. Glycemia ≥ 5.6 mmol/l and < 6.9 mmol/l

Exclusion Criteria:

Subjects with malignant and other acute and chronic infectious and non-infectious disease requiring active pharmacotherapy.

Subjects with with insulin dependent diabetes mellitus or subjects with insulin independent diabetes mellitus taking oral hypoglycemic therapy Subjects with uncontrolled chronic cardiovascular, endocrine, autoimmune, psychiatric, and autoimmune diseases or other condition based on the investigator judgement.

Non adherent subject Systematic use of corticosteroids Pregnant or lactating women Chronic use of supplements (omega 3 unsaturated acids, silymarin, mineral-vitamin supplements) Participation in any other interventional study

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-12-20 (Estimated); Study Completion 2024-08-20 (Estimated)

PRIMARY OUTCOMES:
Change in oxidative stress biomarkers levels: lipid peroxidation index, nitric oxide metabolites, hydrogen peroxide (H2O2), superoxide anion radical (O2-), and glutation (GSH), catalasis(CAT) and superoxid dismutasis(SOD). | From Baseline and after 8 weeks
  ELISA assey
Change in proinflammatori parametars:interleukin-6 (IL-6), tumor necrosis factor-α (TNF- α), high sensitive CRP (hsCRP), leptin, resistin ,vaspin, chemerin ,lipokalin -2 and katepsin | From Baseline and after 8 weeks
  ELISA assey
Change in antiinflammatori parametars:interleukin -5 (IL-5) ,interleukin-10(IL-10), interleukin-12 (IL-12) ,adiponectin and omentin | From Baseline and after 8 weeks
  ELISA assey

SECONDARY OUTCOMES:
Change in inflammation marker level : high sensitivity CRP Turbid mertic test | From Baseline and after 8 weeks
  Turbid metric test
Change in total choleterol (TC), low -density lipoprotein ( LDL), high-density lipoprotein (HDL) and trglicerides Turbid mertic test | From Baseline,after 4 and 8 weeks
  Clinical biochemistry (colorimetric) test and results will be expressed in mmol/l
Change in serum levels homocystein | From Baseline,after 4 and 8 weeks
  Detection by fluoroscence polarization immunoassay
Change in serum levels of vitamin B6-piridoxin ,vitamin B9-folic acid ,vitamin B12-cianocobalamin | From Baseline, after 4 and 8 weeks
  Microparticle enzyme immunoassey
Change in serum levels of glycemia, insulinemia | From Baseline,after 4 and after 8 weeks
  glycemia-hexokinase method,insulinemia-ultrasensitivity test,immunoenzyme test:"sandwich"
Change in serum levels of liver function tests | From Baseline,after 4 and after 8 weeks
  IFCC,reference method with pyridoxyl phosphate
Change in body weight | From Baseline and after 8 weeks
  weight ( kg)
Change in systolic and diastolic blood presure | From Baseline and after 8 weeks
  mm/HG

CONTACTS AND LOCATIONS:
Overall Officials: Ranko Škrbić, Professor, Study Chair — University of Banja Luka
Locations (1):
- Public Health Institution Dom zdravlja Banja Luka, Banja Luka, Republika Srpska, Bosnia and Herzegovina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grabez M, Skrbic R, Stojiljkovic MP, Vucic V, Rudic Grujic V, Jakovljevic V, Djuric DM, Surucic R, Savikin K, Bigovic D, Vasiljevic N. A prospective, randomized, double-blind, placebo-controlled trial of polyphenols on the outcomes of inflammatory factors and oxidative stress in patients with type 2 diabetes mellitus. Rev Cardiovasc Med. 2022 Feb 11;23(2):57. doi: 10.31083/j.rcm2302057. PMID 35229548